CLINICAL TRIAL: NCT02004587
Title: A Single-center, Open-label Trial, Investigating the Pharmacokinetics, Pharmacodynamics and the Safety Profile After a Single Oral Dose of Gemigliptin (Investigational Product) in Healthy Subjects and Subjects With Mild or Moderate Hepatic Impairment and After Multiple Oral Dose in Healthy Subjects
Brief Title: Influence of Hepatic Impairment on Pharmacokinetic (PK) and Pharmacodynamic (PD) of Gemigliptin PK and PD After Multiple Oral Doses in Healthy White Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-DPCL014
Record Dates: First submitted 2013-11-11; First posted 2013-12-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; Pharmacokinetics; Pharmacodynamics; Gemigliptin
MeSH Terms: interventions — LC15-0444

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild hepatic impairment group (Experimental): Mild hepatic impairment group by Child-Pugh scores
  Interventions: Drug: Gemigliptin
- Moderate hepatic impairment group (Experimental): Moderate hepatic impairment group by Child-Pugh scores
  Interventions: Drug: Gemigliptin
- Healthy volunteers (Active Comparator): Gemigliptin dosing in Healthy subjects
  Interventions: Drug: Gemigliptin

INTERVENTIONS:
Drug: Gemigliptin — Gemigliptin is administered to each hepatic impairment subject for single oral dose. Also it is administered to healthy volunteer for single and multiple doses.
  Other Names: Zemiglo

SUMMARY:
The trial will investigate the influence of hepatic function on the PK of gemigliptin. In an additional treatment period, the PK and safety of multiple dosing of gemigliptin in healthy White subjects will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who are able to understand and follow instructions during the study and available for study participation.
* Signed informed consent.
* White

Exclusion Criteria:

* Unwilling or unable to give informed consent.
* As a result of the medical screening process, a study physician considers the subject unfit for the study.
* The subject has a history of drug or other allergy which contraindicated study participation.
* Female subjects who are pregnant or lactating.
* Any other condition (surgical or medical) or history of severe disease with sequelae which increases the risk to the subject or affected absorption, distribution, metabolism or excretion of the study drug or otherwise

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
AUC | Several time points until 72hr
  Blood samples will be prepared at planed points.

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services, Kiel, Schleswig-Holstein, Germany